CLINICAL TRIAL: NCT01007370
Title: Comparison of LMA-Fastrach and I-gel for Blind Tracheal Intubation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NM 2010-001
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: General Anesthesia
Keywords: tracheal intubation; supraglottic airway devices
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LMA-Fastrach (Active Comparator): * Induction of general anesthesia with 1,5-2,5 mg/kg propofol and 1-3 mcg/kg fentanyl and neuromuscular relaxation with 0,6 mg/kg of rocuronium.
  * Direct laryngoscopy, evaluation of laryngeal view grade according to Cormack-Lehane classification
  * Insertion of LMA-Fastrach (sizes 3,4 or 5), establishment of ventilation
  * Evaluation of glottic view through LMA-Fastrach using fibrescope (one out of ten patients)
  * Tracheal intubation through the LMA-Fastrach
  * With the endotracheal tube in place, the anaesthesiologist will proceed to the removal of supraglottic device
  Interventions: Procedure: Tracheal intubation
- I-gel (Active Comparator): * Induction of general anesthesia with 1,5-2,5 mg/kg propofol and 1-3 mcg/kg fentanyl and neuromuscular relaxation with 0,6 mg/kg of rocuronium.
  * Direct laryngoscopy, evaluation of laryngeal view grade according to Cormack-Lehane classification
  * Insertion of I-gel (sizes 3,4 or 5), establishment of ventilation
  * Evaluation of glottic view through I-gel using fibrescope (one out of ten patients)
  * Tracheal intubation through the I-gel
  * With the endotracheal tube in place, the anaesthesiologist will proceed to the removal of supraglottic device
  Interventions: Procedure: Tracheal intubation

INTERVENTIONS:
Procedure: Tracheal intubation — Tracheal intubation through a supraglottic airway device(LMA-Fastrach).
  Arms: LMA-Fastrach
Procedure: Tracheal intubation — Tracheal intubation through a supraglottic airway device(I-gel).
  Arms: I-gel

SUMMARY:
The investigators aim to compare two different types of supraglottic devices for tracheal intubation in patients undergoing elective surgery under general anesthesia.

Our hypothesis is that the use of the I-gel supraglottic airway will result in a higher first attempt success rate of blind tracheal intubation.

DETAILED DESCRIPTION:
Supraglottic airway devices such as LMA-Fastrach and I-gel provide patent airways during general anesthesia.

The LMA-Fastrach is designed to provide a conduit for blind or fiberoptically guided tracheal intubations. However, the success rate of tracheal intubation on the first attempt through this device varies between 50 and 87%.

The I-gel is a newer device for airway management which, with its wide bore, allows direct passage of a tracheal tube. Recent studies suggest that the I-gel is easy to insert and that limited experience is needed before a high success insertion rate is obtained.

In this prospective and randomized study, we will evaluate the performance of both devices for tracheal intubation in patients undergoing elective surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* ASA physical status 1-3
* Patients undergoing elective surgery under general anesthesia, requiring endotracheal intubation

Exclusion Criteria:

* ASA physical status 4-5
* Contraindications to muscle relaxation
* Anticipated or known difficult intubation or ventilation
* Patients with limited mouth opening (less than 2 cm)
* Patients at increased risk of aspiration, or having an history of symptomatic gastroesophageal reflux or hiatal hernia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
First attempt success rate of tracheal intubation. | After successful insertion of tracheal tube

SECONDARY OUTCOMES:
Time needed for successful insertion of a supraglottic device. | After insertion
First and total attempt success rate of supraglottic device insertion. | After insertion
Total time and number of attempts needed to obtain successful tracheal intubation. | After tracheal intubation
Fiberoptic view following the supraglottic device insertion. | After insertion of the device

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Massicotte, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal-Hôpital Notre-Dame, Montreal, Quebec, Canada